CLINICAL TRIAL: NCT06997757
Title: Mobile Health on Improving Efficacy of Plaque Control in Antenatal Women With Gingivitis : A Randomized Controlled Clinical Trial
Brief Title: Mobile Health on Improving Efficacy of Plaque Control in Antenatal Women With Gingivitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: shefaliperiopgids
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Gingivitis
Keywords: mobile health
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOBILE HEALTH (Experimental): Patients will be given Phase I Therapy including Supragingival and Subgingival scaling along with chairside oral hygiene instructions and a mobile phone message reminder will be sent atleast twice a week
  Interventions: Behavioral: Mobile health; Procedure: Phase I Therapy
- CONVENTIONAL THERAPY (Active Comparator): Patients will be given Phase I Therapy including Supragingival and Subgingival Scaling along with chairside oral hygiene instructions
  Interventions: Procedure: Phase I Therapy

INTERVENTIONS:
Behavioral: Mobile health — Instructions for brushing twice daily and using interdental cleaning aids via regular mobile phone messages will be sent atleast twice a week.
  Arms: MOBILE HEALTH
Procedure: Phase I Therapy — Instructions for brushing twice daily and using interdental cleaning aids during appointment only.

SUMMARY:
Oral health education, behavioral therapy and counselling to improve home care in pregnant females along with periodontal therapy can be helpful in treating pregnancy associated gingivitis and pregnancy outcomes

DETAILED DESCRIPTION:
Pregnancy gingivitis has been extensively documented in the previous literature with prevalence of 36-100%. It has been reported that gingivitis is clinically seen in all the pregnant women with increase in gingival changes from 2nd to 8th month of gestation and decreasing in 9th month and post childbirth. The heightened inflammatory response of gingiva towards local irritants is believed to be responsible for the pregnancy gingivitis and has been correlated with the dose-dependent influence of female sex hormones during pregnancy. It has been suggested the increased levels of progesterone exert changes in the microvascular system of gingiva which may aggravate gingivitis. Change in the hormonal level during pregnancy have been found to be predisposing a factor for periodontal changes while Plaque acts as a precipitating factor for pathologic changes.All individuals develop gingivitis in absence of all oral hygiene measures and in healthy individuals a meticulous regime of daily plaque removal can prevent and cure the gingivitis. Since gingivitis is reversible there is a common misconception that a prolonged state of gingival inflammation during pregnancy causes no harm. It causes patient discomfort while brushing and its severity continues to increase during pregnancy. The potential for bacteremia and increased levels of pro-inflammatory cytokines may make effective treatment of gingivitis during pregnancy important for overall maternal and fetal health. In women having pregnancy associated gingivitis, who received periodontal therapy before 28weeks of gestation reported less incidence of Pre-term Labour and Low Birth Weight as compared to women who didn't receive any therapy. Therefore, oral health education, behavioural and counselling to improve home care in pregnant females along with periodontal therapy can be helpful in treating pregnancy associated gingivitis and pregnancy outcomes. Mobile Health is defined by WHO as "a term used for medical and publication health practice supported by mobile devices, such as mobile phones, patient monitoring devices, Personal Digital Assistants (PDAs), and other wireless devices." India has 1.15 billion mobile phone subscribers with 625 million urban & 524 million rural subscribers. India also has the second highest mobile phone connectivity in the world which makes the use of Mobile health in healthcare ideal. Mobile Health can be an effective and valuable treatment as it offers real-time communication between patient and doctor. Mobile health has shown promising results in the medical field Mobile health applications have been found to be an effective adjunctive intervention in self -management by patients with type 2 diabetes. Use of mHealth as an adjunct component in managing gingivitis and in improving daily self-performed oral hygiene has been documented in previous literature.

Research shows that regular prompts and reminders effectively promote and reinforce healthy habits. The average time to form a habit is 66 days with the range of (18- 254days). Improvement in performing oral hygiene has been seen in periodontal patients due to repetition and reinforcement of oral hygiene instructions. It has been documented that text messages are effective in promoting behavioural changes in chronic diseases. Text messages play a key role in encouraging behavioural change and improving health knowledge by offering guidance, warnings, reminders, positive reinforcement and feedback.

Text messaging has been proven in the prevention and management of weight loss, smoking cessation and diabetes. Study has reported higher satisfaction levels among pregnant women who received text messages about prenatal care than those who only received standard prenatal care.

So, in the view of current literature we hypothesise that mobile health reinforcements can contribute to improve oral hygiene behaviours in antenatal women with gingivitis which may have long term benefits postnatally and can improve the pregnancy outcomes. To the best of our knowledge, no study till date has been conducted assessing the effectiveness of Mobile Health in pregnant women diagnosed with gingivitis in improving their oral hygiene after nonsurgical periodontal therapy. So this Randomised controlled Clinical Trial aims to clinically evaluate the effectiveness of Mobile Health in antenatal women with gingivitis in improving efficacy of Plaque control after non surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically Healthy pregnant women of age 18-35 years
2. 8-24 weeks of Gestation
3. Generalized gingivitis (BOP score >30%s, without attachment loss and radiographic bone loss, PPD≤3mm)
4. Access to mobile phone
5. At least 20 natural teeth present

Exclusion Criteria:

1. Presence of systemic diseases that could influence the outcome of periodontal therapy (Diabetes mellitus, Hypertension)
2. Smoking/alcohol consumption
3. Patient currently on any antibiotic therapy
4. Risk for Preterm Birth (Delivery < 37 weeks of gestation)
5. History of periodontal treatment in the last 6 months
6. Physically and mentally impaired patients

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Changes in the Plaque Index will be measured at baseline, 1 month follow up and at 3 month follow up. | 3 months
  Plaque Index as follows will be used for assessment of Plaque :- SCORE 0 : No Plaque SCORE 1: A film of plaque adhering to free gingival margin and adjacent area of the tooth recognized by running a probe SCORE 2 : Moderate accumulation of soft deposits within the gingival pockets or the tooth and gingival margin, which can be seen with naked eyes SCORE 3: Abundance of soft tissue matter on tooth surface and /or gingival margin
Changes in the Gingival Index will be measured at baseline, 1 month follow up and at 3 month follow up | 3 months
  Gingival Index by as follows will be used to assess severity of gingival inflammation:-
  SCORE 0 : Absence of inflammation SCORE 1: Mild inflammation SCORE 2 : Moderate inflammation SCORE 3: Severe inflammation
Changes in the Bleeding on Probing will be measured at baseline, 1 month follow up and at 3 month follow up | 3 months
  It will be measured by walking the periodontal probe at six sites of each tooth, it will be recorded as :
  1- present , if it occurred within 15 seconds of probing 0- absent , if no bleeding occurred It will be calculated in %. After adding all the scores , total score will be divided by the total no. of surfaces assessed and multiplied by 100.
  It will be reported as % sites with bleeding on probing.

SECONDARY OUTCOMES:
Changes in the Probing Pocket Depth will be measured at baseline, 1 month and 3 month follow up | 3 months
  Probing Pocket Depth will be measured as the distance from gingival margin to the base of the pocket .The Probing Depth measurements will be assessed using the periodontal probe. Measurements will be rounded to the nearest whole millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nishi Tanwar, MDS, Principal Investigator — PGIDS , Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No